CLINICAL TRIAL: NCT06067945
Title: Comparison of Marginal Fit and Internal Adaptation in All-Metal Crowns: an in Vitro Experimental Trial
Status: Recruiting | Type: Observational
Sponsor: Altamash Institute of Dental Medicine (Other)
Responsible Party: Principal Investigator, Tooba Shabbir, Post Graduate Trainee, Altamash Institute of Dental Medicine
Other Study IDs: Tshabbir92 Altamash
Record Dates: First submitted 2023-09-25; First posted 2023-10-05 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Evaluation of Marginal and Internal Fit of Metal Crowns

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- NP is given to the non polished group which is group 2: Out of two groups, group 2 is a test group to which rough preparations are assigned
  Interventions: Other: microleakage

INTERVENTIONS:
Other: microleakage — prevention of microleakage and secondary carries

SUMMARY:
The goal of this in vitro study is to compare the marginal fit and internal adaptation of all-metal crowns in polished crown preparations and non-polished crown preparations The main question it aims to answer is: are the non polished tooth preparations comparable to polished preparations? We will compare polish and non polish groups and see their effects on marginal fit and internal adaptation of all metal crown

ELIGIBILITY:
Inclusion Criteria:

1. Phantom teeth
2. Maxillary molars
3. Metal crowns with conventional lost-wax technique for crown fabrication

Exclusion Criteria:

1. Over prepared or underprepared crowns
2. Defective metal crowns
3. Ruptured silicone films upon removal
4. Defective die stone casts

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The phantom teeth (Nissin dental products Inc. Kyoto 601-8469,Japan) will be fixed in the model plaster block type II (Super national, Karachi Pakistan) with full crown and only 2mm of root portion
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
marginal fit | six months
  The margins of fixed restorations refers to the junction between the prepared tooth structure and the crown restoration

SECONDARY OUTCOMES:
Internal fit | six months
  Internal fit is defined as the perpendicular distance between the framework and abutment teeth and the misfit is measured from occlusal/incisal and axial surfaces to the coping

CONTACTS AND LOCATIONS:
Overall Officials: Naseer Ahmad, Ph.D, Study Director — Altamash Institute of Dental Medicine
Locations (1):
- Altamash Institute Of Dental Medicine, Karachi, Sindh, Pakistan